CLINICAL TRIAL: NCT07137416
Title: Phase 1b Study of Pidnarulex and Trastuzumab Deruxtecan in Patients With HER2 Expressing Solid Tumors
Brief Title: Testing the Safety of the Combination of Anti-Cancer Drugs CX-5461 (Pidnarulex) and Trastuzumab Deruxtecan (T-DXd) for Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Solid Tumors and Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-05844; NCI-2025-05844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10720 (Other: Dana-Farber - Harvard Cancer Center LAO); 10720 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2025-08-19; First posted 2025-08-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Invasive Breast Carcinoma; Locally Advanced Breast Carcinoma; Metastatic Breast Carcinoma; Metastatic HER2-Low Breast Carcinoma; Metastatic HER2-Positive Breast Carcinoma; Metastatic Hormone Receptor-Positive Breast Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Triple-Negative Breast Carcinoma; Unresectable Breast Carcinoma; Unresectable HER2-Low Breast Carcinoma; Unresectable HER2-Positive Breast Carcinoma; Unresectable Hormone Receptor-Positive Breast Carcinoma; Unresectable Malignant Solid Neoplasm; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; CX 5461; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Pidnarulex, T-DXd) (Experimental): Patients receive pidnarulex IV over 60 minutes on day 8 of each cycle and T-DXd IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO or MUGA, collection of blood samples, and radiologic imaging throughout the trial. Patients may also undergo biopsy throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Pidnarulex; Procedure: Radiologic Imaging Procedure; Biological: Trastuzumab Deruxtecan

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Pidnarulex — Given IV
  Other Names: CX-5461; CX5461; Pol I Inhibitor CX5461; RNA Pol I Inhibitor CX5461
Procedure: Radiologic Imaging Procedure — Undergo radiologic imaging
Biological: Trastuzumab Deruxtecan — Given IV
  Other Names: DS-8201; DS-8201a; Enhertu; Fam-trastuzumab Deruxtecan-nxki; T-DXd; WHO 10516

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of pidnarulex in combination with trastuzumab deruxtecan in treating patients with breast cancer and other solid tumors that express varying levels of a protein called HER2 and that has spread from where it first started (primary site) to other places in the body (metastatic), that cannot be removed by surgery (unresectable), or that has spread to nearby tissue or lymph nodes (locally advanced). Pidnarulex is an enzyme inhibitor that causes cell death and prevents tumor cell growth. Trastuzumab deruxtecan is in a class of medications called antibody-drug conjugates. It is composed of a monoclonal antibody, called trastuzumab, linked to a chemotherapy drug, called deruxtecan. Trastuzumab attaches to HER2 positive tumor cells in a targeted way and delivers deruxtecan to kill them. Giving pidnarulex in combination with trastuzumab deruxtecan may be safe, tolerable and/or effective in treating patients with metastatic, unresectable, or locally advanced HER2-expressing breast cancer or other solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of CX-5461 (pidnarulex) when used in combination with trastuzumab deruxtecan (T-DXd) in patients with human epidermal growth factor receptor 2 (HER2)-low breast cancer, hormone receptor (HR)-positive HER2-ultralow breast cancer or HER2-positive (immunohistochemistry [IHC] 3+) solid tumors. (Dose escalation primary objective) II. To evaluate safety and tolerability of the combination of CX-5461 (pidnarulex) with T-DXd at the RP2D in patients with HER2-low breast cancer and HR-positive HER2-ultralow breast cancer. (Dose expansion primary objective)

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the plasma pharmacokinetic (PK) profiles of CX-5461 (pidnarulex) and T-DXd when administered in combination.

III. To determine markers of deoxyribonucleic acid (DNA) damage response (DDR) in tumor specimens at baseline and on-treatment in patients with HER2-low and ultralow breast cancer in the dose expansion cohort (pharmacodynamic [PD] objective).

OUTLINE: This is a dose-escalation study of pidnarulex followed by a dose-expansion study.

Patients receive pidnarulex intravenously (IV) over 60 minutes on day 8 of each cycle and T-DXd IV over 30-90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA), collection of blood samples, and radiologic imaging throughout the trial. Patients may also undergo biopsy throughout the trial.

After completion of study treatment, patients are followed up at 30 days and then for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* DOSE ESCALATION PHASE ONLY: Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* DOSE EXPANSION PHASE ONLY: Participants must have histologically or cytologically confirmed invasive breast cancer, with either locally advanced or metastatic disease
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of CX-5461 (pidnarulex) in combination with T-DXd in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count (ANC) ≥ 1,500/mcL

  * No administration of granulocyte colony-stimulating factor (G-CSF) is allowed within 1 week prior to screening assessment
* Platelets ≥ 100,000/mcL

  * No transfusions with red blood cells or platelets are allowed within 1 week prior to screening assessment
* Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN) (or ≤ 2 × institutional ULN in patients with documented Gilbert's syndrome)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 × institutional ULN (or ≤ 5 × ULN in patients with liver metastases)
* International normalized ratio (INR)/prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
* Glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m^2 (using the Cockcroft-Gault equation for participants with creatinine levels above institutional ULN)
* Patients must have had at least one prior line of cytotoxic chemotherapy. Patients can have received an unlimited number of additional lines of chemotherapy, targeted therapy, biologic therapy, or hormonal therapy. Patients must not have progressed on a prior anthracycline in the metastatic setting. Receipt of anthracycline in the (neo)adjuvant setting is allowed, provided that disease recurrence occurred later than 6 months after the completion of treatment
* Prior poly (ADP-ribose) polymerase (PARP) inhibition is allowed
* No specific germline mutation is required
* DOSE ESCALATION PHASE ONLY:

  * HER2-positive (IHC 3+) solid cancers,
  * HR+ HER2 positive/low/ultralow breast cancer or triple negative breast cancer (TNBC) HER2-low breast cancer, with HER2 positive defined by the current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines,
  * HER2-low, with HER2-low defined as IHC 2+/in situ hybridization (ISH)-, IHC 1+/ISH-, or IHC 1+/ISH untested
* DOSE EXPANSION PHASE ONLY:

  * Either the primary invasive tumor and/or the metastasis must be:

    * HER2-low, with HER2-low defined as IHC 2+/ISH-, IHC 1+/ISH-, or IHC 1+/ISH untested. Any estrogen receptor (ER) and progesterone receptor (PR) expression is permitted but must be known, or
    * HR+ HER2-ultralow defined as IHC 0 with membrane staining
* Participants must have at least one lesion that is not within a previously radiated field that is measurable per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Bone lesions are not considered measurable by definition. Biopsy of the lesion that will be used for disease evaluation (measurable disease) is not allowed in the dose expansion portion of this study
* Peripheral neuropathy grade ≤ 1
* Patients must have left ventricular ejection fraction (LVEF) ≥ 50% by either an echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within 28 days before randomization/enrollment
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of CX-5461 (pidnarulex) and T-DXd on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) 14 days prior to study entry and for the duration of study participation and for at least 7 months (women of childbearing potential [WOCBP] only) after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women should not breastfeed while taking CX-5461 (pidnarulex) and T-DXd and for 7 months after cessation of treatment. Men treated or enrolled on this protocol must also agree to use adequate contraception 14 days prior to the study, for the duration of study participation, and 6 months after completion of CX-5461 (pidnarulex) and T-DXd administration
* Women of non-child-bearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases, a blood sample with simultaneous follicle-stimulating hormone [FSH] > 40 mIU/mL and estradiol < 40 pg/mL [< 147 pmol/L] is confirmatory) or on ovarian suppression are eligible. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Male patients must not freeze or donate sperm starting at screening and throughout the study period, and at least 6 months after the final study drug administration. Preservation of sperm should be considered prior to enrollment in this study
* Female patients must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives (LAR) may sign and give informed consent on behalf of study participants
* Patients who have had chest radiation therapy within 4 weeks (2 weeks for palliative stereotactic radiation therapy). These patients will be excluded because T-DXd is known to increase the risk of developing pneumonitis

Exclusion Criteria:

* Patients with a history of (non-infectious) interstitial lung disease (ILD) that required steroids, have current ILD, or where there is suspected ILD that cannot be ruled out by imaging at screening. These patients will be excluded because T-DXd is known to increase the risk of developing ILD and pneumonitis
* Patients with clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within three months of the study enrollment, severe asthma, severe chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, etc.), and any autoimmune, connective tissue or inflammatory disorders with potential pulmonary involvement (i.e., Rheumatoid arthritis, Sjogren's, sarcoidosis, etc.), or prior pneumonectomy at the time of screening. These patients will be excluded because T-DXd is known to increase the risk of developing ILD and pneumonitis
* Patients who have had chemotherapy (including antibody drug therapy, retinoid therapy, hormonal therapy for cancer) within 3 weeks (2 weeks or five half-lives, whichever is longer for small-molecule targeted agents such as 5-fluorouracil-based agents, folinate agents), weekly paclitaxel; 6 weeks for nitrosoureas or mitomycin C. These patients will be excluded to allow for recovery of toxicities related to chemotherapy and minimize risk of drug interactions
* Patients who have had cancer immunotherapy including monoclonal antibody therapy within 4 weeks
* Patients who have had a major surgery within 4 weeks
* Patients with unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to grade ≤ 1 or baseline. Patients with chronic grade 2 toxicities may be eligible (e.g., grade 2 chemotherapy-induced neuropathy). Patients should no longer be symptomatic nor require treatment with corticosteroids or anticonvulsants and must have recovered from the acute toxic effect of radiotherapy
* Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity of CX-5461 (pidnarulex) will be determined based on their potential to interact with the CYP3A4 isozyme. Specifically, subjects taking strong CYP3A4 inhibitors or strong CYP3A4 inducers will be excluded from participation in the trial. A list of agents that interact with CYP450 isoenzymes is provided
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CX-5461 (pidnarulex), T-DXd, or the inactive ingredients in the drug products, including patients who have a history of severe hypersensitivity reactions to other monoclonal antibodies
* Patients with a corrected QT interval (QTc) prolongation to > 470 ms (females) or > 450 ms (males) based on average of the screening triplicate 12-lead electrocardiogram (ECG)
* Patients with clinically significant corneal disease, cicatricial conjunctivitis or active ocular surface disease in the opinion of the investigator
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous
* Pregnant women are excluded from this study because CX-5461 (pidnarulex) and T-DXd are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with CX-5461 (pidnarulex) and T-DXd, breastfeeding should be discontinued if the mother is treated with CX-5461 (pidnarulex) and T-DXd and avoided for 7 months after the last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-10-05 (Estimated); Primary Completion 2028-01-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (dose escalation phase) | Up to completion of dose-escalation
  The dose escalation will follow a Bayesian Optimal Interval design with a target dose limiting toxicity rate of 25%.
Incidence of adverse events with drug combination at the recommended phase 2 dose (dose expansion phase) | Up to 3 years

SECONDARY OUTCOMES:
Tumor response rate | Up to 3 years
  Radiological response will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1 criteria and will be graded as complete response (CR), partial response (PR), stable disease (SD), and progressive disease. Response rate (CR + PR) and clinical benefit rate (CR + PR + SD > 24 weeks) will be summarized by frequencies and percentages, by dose level.
Plasma concentrations of CX-5461 (pidnarulex) and trastuzumab deruxtecan | Cycle (C) 1 day (D) 1, C1D8, C1D10, C1D15, C2D1, C2D8, C2D10, C2D15 (cycle length = 21 days)
  Will measure the plasma concentrations of both CX-5461 (pidnarulex) and deruxtecan over time. Area under the curve, maximum concentration, time to reach maximum concentration, and elimination half-life will be calculated for the two study drugs and summarized by dose level.
Markers of deoxyribonucleic acid (DNA) damage repair (DDR) | At baseline and on-treatment
  The secondary, pharmacodynamic endpoint is to determine markers of DDR in tumor specimens at baseline and on-treatment in patients with advanced HER2-low breast cancer in the dose expansion. For the DDR assay, levels exceeding 4% nuclear area positive (NAP) γH2AX, 4% NAP pNBS1, and 5% cells with ≥ 5 Rad51 nuclear foci indicate a DNA damage activation response.

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Lynce, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (1):
- Dana-Farber - Harvard Cancer Center LAO, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm